CLINICAL TRIAL: NCT01364675
Title: Primary Prevention of Cardiovascular Disease in Pre-diabetic & Pre-hypertensive Subjects Using Multiple Risks Reduction Strategy: A Multi-center, Double-blind, Randomized Controlled Trial
Brief Title: Primary Prevention of Cardiovascular Disease (CVD) in Pre-diabetic & Pre-hypertensive Subjects
Acronym: PPCVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Ubon Ratchathani Public Health Office, Thailand (Other Government); National Health Security Office, Thailand (Other); The Government Pharmaceutical Organization (Other Government)
Responsible Party: Phisitt Vejakama, Section for clinical epidemiology, Faculty of medicine, Ramathibodi hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12011
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Pre-diabetes; Pre-hypertension
Keywords: Impaired fasting glucose; Impaired glucose tolerance; Pre-diabetes; Pre-hypertensives; Cardiovascular events
MeSH Terms: conditions — Glucose Intolerance; Prehypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin+Enalapril+Simvastatin (Experimental)
  Interventions: Drug: Metformin+Enalapril+Simvastatin
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Metformin+Enalapril+Simvastatin — Poly-pill - composed of Metformin (500 mg), Enalapril (10 mg) and Simvastatin (10 mg) in single tablet given once daily after dinner for 4 years
  Other Names: Poly-pill
  Arms: Metformin+Enalapril+Simvastatin
Drug: Placebo tablet — Identical Placebo Tablet
  Other Names: Placebo
  Arms: Placebo tablet

SUMMARY:
The purpose of this study is to determine whether treating pre-diabetic & pre-hypertensive individuals using multiple drugs intervention (anti-hypertensive drugs (i.e., ACEI) plus anti-glycemic drug (i.e., metformin) plus anti-hyperlipidemic drug (statin)) would lower Cardiovascular Disease (CVD) events.

DETAILED DESCRIPTION:
The risks of CVD are not confined to a subset of established "hypertensive" or "diabetic" population, but also increase among those with suboptimal blood pressure and glycemic level, namely "pre-hypertensive" or "pre-diabetic" population. Evidence on the effectiveness of drug interventions to lower CVD events in pre-clinical stage population has been scant.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes
* Pre-hypertensives
* LDL-Cholesterol >= 100 < 190 mg/dl
* BMI >= 23
* Estimated GFR >= 60 ml/min/1.73 m2 (MDRD equation)
* Willing to participate and provide written inform consent

Exclusion Criteria:

* Current involved in other studied medications
* Regular use of corticosteroids
* Current use of weight loss medication
* History of renal disease
* Active liver disease including jaundice, chronic hepatitis with ALT >= 2.5 the upper normal limit
* Active malignancy
* Major psychiatric disorder
* Diseases and medications that affect glucose tolerance (e.g. pheochromocytoma, Cushing's syndrome, acromegaly, steroid-dependent asthma, protease inhibitors, antipsychotics)
* Nursing women, pregnant women, or those that plan to become pregnant in the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8900 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Events | 4-year
  Fatal or Non-fatal Myocardial Infarction, Angina Pectoris, Congestive Heart Failure, Coronary Revascularization, Fatal or Non-fatal Stroke, Amputation of Lower Extremities (non-traumatic cause)

SECONDARY OUTCOMES:
Micro-vascular Complications | 4-year
  Renal dysfunction, ESRD (on dialysis or kidney transplantation), Progression of Albuminuria, Retinopathy
Cumulative Incidence of Diabetes | 4-year
Cumulative Incidence of Hypertension | 4-year
Incidence of Individual Cardiovascular Disease | 4-year
  Coronary Artery Disease - Myocardial Infarction, Angina Pectoris, Congestive Heart Failure, Coronary Revascularization
  Stroke- Cerebral Hemorrhage, Cerebral Infarction, Subarachnoid Hemorrhage
  Peripheral Artery Disease- Leg amputation, endovascular or surgical intervention in leg arteries

CONTACTS AND LOCATIONS:
Overall Officials: Phisitt Vejakama, M.D., Principal Investigator — Section for clinical epidemiology and bioststistics, Faculty of medicine, Ramathibodi hospital
Locations (1):
- Ubon ratchathani Public Health Office, Muang District, Changwat Ubon Ratchathani, Thailand